CLINICAL TRIAL: NCT04563767
Title: Feasibility of Utilizing the Infinitome Program to Evaluate Abnormal Large Scale Brain Networks in Alzheimer's Disease
Brief Title: Feasibility - Infinitome
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A20-199
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infinitome: All patients will be in the same cohort. No intervention will be administered. Patients will undergo a structural magnetic resonance imaging (MRI) as part of their standard of care. Added on will be the resting state fMRI (rs-fMRI). The rs-fMRI data will be analyzed.
  Interventions: Procedure: Infinitome

INTERVENTIONS:
Procedure: Infinitome — Added sequence of rs-fMRI.

SUMMARY:
The Infinitome Program from Omniscient has the ability to identify abnormal brain networks or connectomes using resting state functional MRI (rs-fMRI). This technology, which visualizes brain networks in three dimensions, was originally developed to ensure neurosurgeons avoid inadvertently lesioning cognitively eloquent brain regions during surgical operations. The potential of Infinitome in identifying connectome dysfunction for neurodegenerative diseases such as Alzheimer's disease has yet to be explored. This diagnostic technique may play a critical role for identifying disease brain networks that may benefit from targeted interventions in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of mild, moderate, or severe Alzheimer's disease
2. Age: 40 - 90 Years
3. Patients who are clinically indicated for an MRI

Exclusion Criteria:

1. fMRI contraindicated (eg. Implantable device, pacemaker, metallic implants, etc.)
2. Subject unable to tolerate sitting for a one hour fMRI
3. Other concerns as determined by the investigator

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HealthPartners Neurology Clinic in Saint Paul, MN undergoing care for Alzheimer's disease.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rosenbloom, MD, Principal Investigator — HealthPartners Neurology
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infinitome
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infinitome
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Rs-fMRI
Description: Percent of subjects who complete the sequence of the fMRI protocol. Range: 0-100. Higher percentage indicates more completion.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Infinitome
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Number of Subjects Whose Images Completed Analysis
Description: Percent of subjects whose images were uploaded and analyzed by the Infinitome program. Range: 0-100. Higher percentage indicates more completion.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Infinitome
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Only observed during MRI.
Arm/Group | Infinitome
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT04563767/Prot_SAP_000.pdf